CLINICAL TRIAL: NCT04721756
Title: A Phase I Study Evaluating the Safety and Imaging Characteristics of 18F-LY3546117 Injection in Subjects Who Are Undergoing Treatment With Immune Checkpoint Inhibitors
Brief Title: Early Clinical Evaluation of 18F-LY3546117 in Tumor Imaging
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-LY3546117-01
Record Dates: First submitted 2021-01-13; First posted 2021-01-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Neoplasms; Neoplasms Malignant
Keywords: Cancer Imaging
MeSH Terms: conditions — Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 18F-LY3546117 Scan Cohort 1 (Experimental): 18F-LY3546117 PET scan at baseline and between 14-42 days after initiation of immune checkpoint therapy
  Interventions: Drug: 18F-LY3546117 Injection; Procedure: PET Scan
- 18F-LY3546117 Scan Cohort 2 (Experimental): 18F-LY3546117 PET scan at time of immune checkpoint therapy response
  Interventions: Drug: 18F-LY3546117 Injection; Procedure: PET Scan

INTERVENTIONS:
Drug: 18F-LY3546117 Injection — 370 megabecquerel (MBq) intravenous injection
Procedure: PET Scan — positron emission tomography (PET) scan

SUMMARY:
Immuno-Oncology (IO) therapies have revolutionized cancer therapy and are becoming the standard of care for many cancers. Monitoring how well IO therapies work against cancer is difficult due to the complexity of the immune system and the fact that an immune response may initially increase, rather than decrease, the size of a tumor. An early response marker would be beneficial to determine which patients should remain on a given treatment or combination of treatments, and which patients should seek other treatment options. 18F-LY3546117 is a radiolabeled tracer that binds to a specific protein (Granzyme B) that is found in the human immune system and is thought to trigger programmed cell death. It is thought that imaging Granzyme B activity in tumors and elsewhere in the body using a Positron Emission Tomography (PET) scan will allow doctors to monitor the progress of IO therapy.

ELIGIBILITY:
Inclusion Criteria (Cohort 1):

* At least one imageable tumor greater than or equal to 15 mm in the longest diameter
* Confirmed diagnosis of cancer with a high likelihood of response to immuno-oncology therapy (melanoma or non-small cell lung cancer, or other malignancies with sponsor approval) and planned mono- or combination therapy with immuno-oncology therapy
* Life expectancy of greater than 6 months

Inclusion Criteria (Cohort 2):

* At least one imageable tumor greater than or equal to 15 mm in the longest diameter or a tumor assessable by PET in the opinion of the radiologist
* Received treatment with an immune checkpoint inhibitor with evidence of response
* Life expectancy of greater than 6 months

Exclusion Criteria:

* Subjects who plan to receive chemotherapy or radiation therapy during study participation
* Prior history of failed immune checkpoint inhibitor therapy
* Subjects who require steroid or other immunosuppressive medications within 2 weeks of the PET scan.
* Females of childbearing potential who are not surgically sterile, not refraining from sexual activity, or not using effective methods of contraception. Females of childbearing potential must not be pregnant or breastfeeding at screening and agree to avoid becoming pregnant for 24 hours following study drug administration.
* Females and males must agree to refrain from sexual activity or to use effective contraceptive methods for 24 hours following study drug administration and during study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Uptake of 18F-LY3546117 in tumor foci and other organs of the body | Day 14 up to Day 42 of immune checkpoint inhibitor therapy
  Visual uptake in the tumor as assessed by sponsor expert reader (Yes/No)
Cohort 2: Uptake of 18F-LY3546117 in tumor foci and other organs of the body | At immune checkpoint inhibitor treatment response (Day 42 up to 6 months post-treatment)
  Visual uptake in the tumor as assessed by sponsor expert reader (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Avid Medical Director, Study Director — Avid Radiopharmaceuticals, Inc.
Locations (1):
- Olivia Newton-John Cancer Institute and Austin Health, Heidelberg, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No